CLINICAL TRIAL: NCT07213531
Title: Enhanced Valves Interventions and Safe AI Generated End Results
Acronym: ENVISAGE
Status: Recruiting | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: Centre Hospitalier Universitaire de Bordeaux, FRANCE (Unknown); Materialise (Industry); Pie Medical Imaging (Unknown); Clinique Pasteur Toulouse (Other); Centre Cardiologique du Nord (Other); CHU Rennes,France (Unknown); San Raffaele University Hospital, Italy (Other); Istituto clinico Città di Brescia (Unknown); Unity Health Toronto (Other); University Hospital, Marseille (Other); Lille University Hospital (Unknown); Hospitaux Universitaires Paris Sud (Unknown); Montefiore Medical Center (Other); University Medical Center Mainz (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Vancouver Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX2024/50
Record Dates: First submitted 2025-09-24; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Heart Valve Disease; TAVI; M-TEER; TTVI; TMVI; T-TEER; Mitraclip; TriClip
Keywords: Medical imaging; CT; Artificial intelligence; M-TEER; T-TEER; TAVI; TMVI; valvulopathy; predictive algorithms
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- TAVI: All patients who have had TAVI with a third generation transcatheter heart valve (THV). Medical imaging data (CT, TEE) and preoperative clinical data will be collected for analysis.
  Interventions: Diagnostic Test: Medical imaging analysis via artificial intelligence algorithms
- TMVI: Patients who have had a TMVI with a dedicated transeptal device and screen failures. Medical imaging data (CT, TEE) and preoperative clinical data will be collected for analysis.
  Interventions: Diagnostic Test: Medical imaging analysis via artificial intelligence algorithms
- TTVI: Patients who have had a TTVI with a dedicated device and screen failures. Medical imaging data (CT, TEE) and preoperative clinical data will be collected for analysis.
  Interventions: Diagnostic Test: Medical imaging analysis via artificial intelligence algorithms
- M-TEER: All patients who have had a M-TEER with 1) G4 or newer iteration of MitraClip or 2) G2 or newer iteration of Pascal. Medical imaging data (CT, TEE) and preoperative clinical data will be collected for analysis.
  Interventions: Diagnostic Test: Medical imaging analysis via artificial intelligence algorithms
- T-TEER: All patients who have had a T-TEER with G4 or newer iteration of TriClip or 2) G2 or newer iteration of Pascal. Medical imaging data (CT, TEE) and preoperative clinical data will be collected for analysis.
  Interventions: Diagnostic Test: Medical imaging analysis via artificial intelligence algorithms

INTERVENTIONS:
Diagnostic Test: Medical imaging analysis via artificial intelligence algorithms — Development of AI algorithms based on pre-procedural imaging annotations and clinical informations to predict the transcatheter procedural outcomes

SUMMARY:
This non-interventional study aims to use artificial intelligence to improve the prediction of transcatheter heart valve interventions and optimize patient outcomes. It is based on the analysis of retrospective data from various specialized centers worldwide.

DETAILED DESCRIPTION:
The ENVISAGE study is a non-interventional, retrospective research study designed to validate an artificial intelligence (AI)-based framework for the automated analysis of cardiac imaging data, including multi-slice cardiac computed tomography (CT) and transesophageal echocardiography (TEE). The primary objective is to predict the success of transcatheter heart valve interventions, including aortic, mitral, and tricuspid valve interventions (TAVI, TMVI, M-TEER, T-TEER). The AI framework developed in this study will rely on deep learning algorithms, particularly convolutional neural networks (CNNs) and other advanced models, to automatically segment critical anatomical structures and perform accurate measurements of these structures from CT and TEE images. These measurements will then be combined with pre-interventional clinical data to optimize patient selection and intervention planning, as well as to predict surgical outcomes with high accuracy. AI will also aim to reduce human error and inter-observer variability in the interpretation of cardiac images, which could significantly improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients who have reached the age of legal majority under local laws.

* For TAVI group: All patients who have had TAVI with a third generation transcatheter heart valve (THV), with an available pre-procedural optimal quality CT scan as defined by an ECG- gating CT with:

  1. five to ten image volumes at cardiac phases from 5% to 95% R-R
  2. 0.625 mm slice thickness
  3. 0.625 mm spacing between slices
  4. 0.88 mm in-plane pixel spacing
* For TMVI group: Patients who have had a TMVI with a dedicated device and screen failures, with an available optimal quality CT scan.
* For TTVI group: Patients who have had a TTVI with a dedicated device and screen failures, with an available optimal quality CT scan.
* For M-TEER: All patient who have had a M-TEER with 1) G4 or newer iteration of MitraClip or 2) G2 or newer iteration of Pascal, with available pre-procedural TEE videos images from one of two vendors: Phillips or GE, with clear identifiable views of the Mitral valve, frame per second equal or higher than 40 frames per second, acceptable 3D reconstructions.
* For T-TEER: All patient who have had a T-TEER with G4 or newer iteration of TriClip or 2) G2 or newer iteration of Pascal, with available pre-procedural TEE videos images from one of two vendors: Phillips or GE, with clear identifiable views of the Tricuspid valve, frame per second equal or higher than 40 frames per second, acceptable transgastric image with acceptable 3D reconstructions.

Exclusion Criteria:

* For TAVI group: Valve-in-valve procedures
* For TMVI group: Valve-in-valve and valve-in-ring procedures
* For TTVI: Valve-in-valve and valve-in-ring procedures
* For M-TEER: G3 or older MitraClip, G1 Pascal
* For T-TEER: G3 Triclip, G1 Pascal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart valve disease eligible for transcatheter interventions (TAVI, M-TEER, TMVI, TTVI).
Sampling Method: Non-Probability Sample
Enrollment: 21000 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Accuracy of transcatheter AI predictions | Preoperative phase: automated segmentation and measurements compared with manual assessments; Postoperative phase at day 30: comparison of predicted results with actual clinical patient outcomes.
  Validation of artificial intelligence algorithms for automatic segmentation of anatomic structures and imaging measurements, and prediction of the success of transcatheter interventions.
  Output of AI algorithm:
  * Sizes, types, and number of devices to be implanted
  * Device success
  * Percentage risk of permanent pacemaker implantation (for TAVI and TTVI)
  * Percentage risk of 30-day (para)valvular regurgitation for TAVI, and residual regurgitation for M-TEER and T-TEER
  * Single leaflet detachment for M-TEER and T-TEER
  * Left ventricular outflow tract obstruction for TMVI.
  Key success indicators:
  * First, independent retrospective validation dataset AI algorithms predict procedural outcome with >90% accuracy and low inter-reader observer variability when compared to measured procedural outcome.
  * Second independent retrospective dataset, perform a study to validate AI algorithms with >90% accuracy and low inter-reader observer variability when compared to measured procedural outcome.

SECONDARY OUTCOMES:
Performance of AI algorithms in CT and TEE image analysis | Through study completion, an average of 2 years (retrospective analysis and validation of algorithms).
  Development and evaluation of AI algorithm training platform for data analysis of patients undergoing transcatheter valve procedures. Comparison of AI model performance with existing benchmarks and manual analyses

OTHER OUTCOMES:
AI-based discovery of clinical knowledge for patient selection | Baseline (pre-procedural) and post-procedural (day 90) analysis
  Comparison of AI's ability to standardize patient selection, treatment planning and clinical outcomes with traditional methods. Assessment of accuracy in predicting patient outcomes and reducing procedure-specific complications.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Modine, MD, PhD, Principal Investigator — University Hospital Bordeaux, France; Walid Ben Ali, MD, PhD, Principal Investigator — Montreal Heart Institute
Locations (15):
- Montefiore Medical Center New York, New York, New York, United States
- Canada (3):
  - Montreal Heart Institute, 5000 Rue Bélanger, Montréal, Montreal, Quebec
  - St Michael's Hospital Toronto, Toronto
  - St Paul's Hospital Vancouver, Vancouver
- France (7):
  - Centre Hospitalier Universitaire (CHU) de Bordeaux, 12 rue Dubernat 33404 Talence cedex, Bourdeaux
  - CHU Lille, Lille
  - CHU Marseille, Marseille
  - Centre Cardiologique du Nord Paris, Paris
  - Institut Cardiovasculaire Paris-Sud Paris, Paris
  - Centre Hospitalier Universitaire Rennes, Rennes
  - Clinque Pasteur Toulouse - France, Toulouse
- Germany (2):
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Heart Valve Center Mainz, Mainz
- Italy (2):
  - Istituto Clinico Città di Brescia, Brescia
  - San Raffaele Heart Valve Center Milan, Milan

IPD SHARING:
Plan to Share IPD: No